CLINICAL TRIAL: NCT01609322
Title: Exposure Therapy for Fear of Falling in Older Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Julie Wetherell, Professor, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R34MH086668 (NIH); R34MH086668 (NIH)
Record Dates: First submitted 2012-05-29; First posted 2012-05-31 (Estimated); Last update posted 2013-12-23 (Estimated); Status verified 2013-12

CONDITIONS: Fear of Falling
Keywords: fear of falling; agoraphobia
MeSH Terms: conditions — Agoraphobia | interventions — Exercise; Educational Status

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Education about falls (Active Comparator): In-person education about falls with a health educator.
  Interventions: Behavioral: Fall prevention education
- Activity, Balance, Learning, and Exposure (Experimental): Intervention combining medication review, exercise, home safety evaluation, and exposure therapy.
  Interventions: Behavioral: Activity, Balance, Learning, and Exposure

INTERVENTIONS:
Behavioral: Activity, Balance, Learning, and Exposure — An in-home intervention that integrates exposure therapy with cognitive restructuring, exercise, and a home safety evaluation.
  Arms: Activity, Balance, Learning, and Exposure
Behavioral: Fall prevention education — In-home, individual sessions with a health educator regarding fall prevention
  Arms: Education about falls

SUMMARY:
This project aims to test the efficacy of an in-home intervention, "Activity, Balance, Learning, and Exposure" (ABLE), which integrates exposure therapy with cognitive restructuring, exercise, and home safety evaluation for older adults with excessive fear of falling. The intervention will be conducted by a licensed physical therapist. A control intervention will be conducted by a health educator. The specific aims of the study are to test the feasibility, acceptability, tolerability, and safety of the ABLE intervention.

DETAILED DESCRIPTION:
Approximately 7-14% of older adults living independently in the community, including more than 5% of those who have never experienced a fall, experience moderate to severe fear of falling. Fear of falling leads to decreased physical activity, disability, loss of independence, depression, anxiety, reduced social engagement, and poor quality of life. It is also a major independent risk factor for falls.

Interventions targeting fear of falling, typically delivered in groups and incorporating cognitive restructuring, education, and exercise, have been shown to increase fall-related self-efficacy. Avoidance is resistant to treatment, however, and more than one-third of patients enrolled in these interventions drop out. Factors associated with attrition include high levels of fear and avoidance, indicating that the individuals most in need of such programs are those most likely to withdraw prematurely. These data suggest that avoidance should be targeted in treatment, and that interventions should be designed to reach very fearful individuals who are most likely to drop out of traditional fear of falling programs.

Participation in this study will last up to 8 months. Participants will be randomly assigned to receive either the ABLE intervention or an education control condition. The control condition will consist of in-person education about falls to control for the time and attention provided in the ABLE arm.

ELIGIBILITY:
Inclusion Criteria:

1. Age 65 years old or older.
2. Severe fear as measured by a brief FES-I score > or = 13.
3. Low to moderate actual risk of falls as set out in Lamb et al. (2008).
4. Distress or functional impairment due to fear of falling.
5. Approval from the patient's primary health care provider.

Exclusion Criteria:

1. Medical condition that would interfere with the safe conduct of the intervention or compromise study participation.
2. Bedbound, wheelchair-dependent, paralyzed in the lower extremities, or requiring the assistance of another person to transfer, walk, or perform intervention exercises within the home.
3. Dementia or cognitive impairment as measured by a score above 10 on the Blessed Orientation Memory Test.
4. Corrected visual acuity < 20/60.
5. Current participation in psychotherapy or professional rehabilitation services (PT, OT) or in the process of being referred or evaluated for such services. Patients who develop a need for such services during their participation will complete an assessment prior to commencing the outside therapy but will be allowed to continue in the study.
6. Active suicidal ideation
7. Lifetime diagnosis of bipolar I or II disorder or any psychotic disorder.
8. Alcohol or other substance abuse or dependence within six months.
9. Psychosocial factors that would compromise study participation (e.g. homelessness, no telephone).
10. History of osteoporotic fracture.
11. Experiencing 3 or more falls in the past year.
12. Body Mass Index of 17.0 or under.
13. Significant orthostasis, defined as a 20 point or greater difference between seated and standing blood pressure, either systolic or diastolic.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-08; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Fear of falling | 2 months (primary)
  Fear of Falling will be measured using the Falls Efficacy Scale - International (FES-I), a version of the most widely used measure of falls self-efficacy. Assessments are performed at baseline, 1 month, 2 months (end of intervention - primary outcome point). We will also collect data at 5 months (3 month follow-up) and 8 months (6 month follow-up).
Activity avoidance | 2 months (primary)
  Activity avoidance will be assessed using a modified version of the Activity Card Sort, a set of photographs of older adults engaged in various activities that is used in rehabilitation settings. Assessments are performed at baseline, 1 month, 2 months (end of intervention - primary outcome point), 5 months (3 month follow-up), and 8 months (6 month follow-up).

SECONDARY OUTCOMES:
Physical activity - self-report | 2 months (primary)
  Self-reported physical activity will be assessed with the Physical Activities Scale for the Elderly (PASE).
Physical activity | 2 months
  Accelerometers will also be used to measure physical activity. Patients in the study will wear an Actigraph battery-operated activity monitor worn around the waist to measure physical activity continuously during waking hours. Assessment will occur before and after the intervention.
Physical Performance | 2 months (primary)
  Physical performance will be measured using the Short Physical Performance Battery (SPPB), which includes measured of balance, walking, and lower body strength.
Quality of Life | 2 months (primary)
  Quality of life will be measured with the Quality of Life Inventory (QOLI).
Depressive and Anxiety symptoms | 2 months (primary)
  Depressive and anxiety symptoms will be assessed with the Hospital Anxiety and Depression Scale (HADS), a 14-item self-report measure with subscales assessing depressive and anxiety symptoms that does not include somatic items such as fatigue that can be associated with aging or medical conditions rather than psychiatric disorders.
Agoraphobic Avoidance | 2 months (primary)
  Agoraphobic avoidance will be measured using the 5-item agoraphobia subscale of the Fear Questionaire (FQ).
Post Traumatic Stress Disorder Symptoms | 2 months (primary)
  Post Traumatic Stress Disorder (PTSD) symptoms will be measured with the 6-item abbreviated form of the PTSD Checklist (PCL).
Fear of Falling | 2 months (primary)
  Fear of falling will be measured using the Falling Questionaire, a 15-item survey assessing attitudes towards falling.
Avoidance | 2 months (primary)
  Avoidance of activities will be measured using the Fear of Falling Avoidance-Behavior Questionaire (FFABQ), a 14-item measure to assess avoidance behaviors.
Falls | 2 months (primary)
  Recorded on fall diaries provided to investigators throughout the 2-month intervention and 6-month follow-up period.

CONTACTS AND LOCATIONS:
Overall Officials: Julie Wetherell, PhD, Principal Investigator — UCSD
Locations (1):
- University of California San Diego, San Diego, California, United States

REFERENCES:
- [Derived] Wetherell JL, Bower ES, Johnson K, Chang DG, Ward SR, Petkus AJ. Integrated Exposure Therapy and Exercise Reduces Fear of Falling and Avoidance in Older Adults: A Randomized Pilot Study. Am J Geriatr Psychiatry. 2018 Aug;26(8):849-859. doi: 10.1016/j.jagp.2018.04.001. Epub 2018 Apr 12. PMID 29754811